CLINICAL TRIAL: NCT03956277
Title: A Single-center, Feasibility Study to Evaluate the Use and Safety of the Percutaneous Ultrasound Gastrostomy Technique
Brief Title: Single-center, Feasibility Study to Evaluate the Use and Safety of the Percutaneous Ultrasound Gastrostomy Technique
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CoapTech (Industry)
Collaborators: University of Maryland, Baltimore (Other); University of Maryland, Baltimore Washington Medical Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1801004
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-01

CONDITIONS: Gastrostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Observational PUG: Patients receive gastrostomy via percutaneous ultrasound gastrostomy.
  Interventions: Device: PUG

INTERVENTIONS:
Device: PUG — This methodology involves using ultrasound to place gastrostomy tube (g-tube itself is off the shelf).

SUMMARY:
This is a single-center, non-randomized, non-blinded feasibility study to evaluate the performance, safety and tolerability of the Percutaneous Ultrasound Gastrostomy (PUG) procedure that utilizes a novel device in conjunction with widely available ultrasound technology. The procedure will be performed in 40eligible subjects. Patients will be followed for 2 days following performance of PUG to assess for potential complications. If the patient remains hospitalized they will be assessed through Day30 for potential complications.

ELIGIBILITY:
Inclusion Criteria:

* •Written informed consent must be obtained before any study-specific assessment is performed •Male or female ≥18 years of age•BMI between 20 and 30•Indication for gastrostomy tube placement determined to be present by the primary clinical care team•Patient determined to be an appropriate candidate for PEG or PUG by the study team•Women of childbearing potential must have negative serum or urine pregnancy test duringthe current hospitalization

Exclusion Criteria:

* •BMI <20 or > 30•Temperature ≥ 38 C •Systolic BP < 100 or > 180 mmHg•Heart Rate < 50 or > 110•Presence of a contraindication to being in proximity to a magnet (e.g. pacemaker).•History of prior gastrostomy or gastrectomy (partial or complete).•Patients with hematocrit <25%, or a history of blood transfusion within the 14 days prior to screening, or active life-threatening GI bleeding. •Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test. •Involvement in other investigational trials within 30 days prior to screening.•Any other medical condition(s) that may putthe patient at risk or influence study results in the investigator's opinion, or that the investigator deems unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who meet the inclusion and exclusion criteria who are indicated for gastrostomy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-10-14 (Estimated); Study Completion 2024-02-04 (Estimated)

PRIMARY OUTCOMES:
Technical Success of PUG | Immediate
  proportion of PUG procedures that result in successful placement of a gastrostomy tube

SECONDARY OUTCOMES:
SAE Rate | 30 days
  compare the rate of serious complications during the immediate procedural period between the PUG placement and a historical cohort of matched controls who underwent gastrostomy placement using the PEG technique.
Complication Rate | 30 days
  compare the rate of other complications during the immediate procedural period between the PUG placement and a historical cohort of matched controls who underwent gastrostomy placement using the PEG technique.

CONTACTS AND LOCATIONS:
Overall Officials: Gentry Wilkerson, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No